CLINICAL TRIAL: NCT04025268
Title: Development of a Group Prenatal Care Intervention to Address Maternal and Child Non-Communicable Disease (NCD) Risk in American Samoa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1609018463
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: 2 cohort double blinded randomized control trial
Who Masked: Participant, Care Provider
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pregnant women receiving group prenatal care (GPNC) (Active Comparator): Overweight/obese pregnant women will be recruited from the prenatal care clinic at the Lyndon B Johnson Tropical Medical Center (LBJTMC) in Pago Pago, American Samoa. These women will be randomized to receive the 10-session GPNC intervention.
  Interventions: Behavioral: Group Prenatal Care (GPNC)
- pregnant women receiving standard of care (SOC) (Active Comparator): Overweight/obese pregnant women will be recruited from the prenatal care clinic at the Lyndon B Johnson Tropical Medical Center (LBJTMC) in Pago Pago, American Samoa. These women will be randomized to continue with standard of care (SOC) prenatal care visits.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Group Prenatal Care (GPNC) — GPNC participants will attend 11 group sessions total: 10 during pregnancy and one postpartum. Each session will be 90-100 minutes long. Groups will collectively identify the preferred time of day for these sessions. Groups of 10 women will be led by a locally trained, Samoan nurse-midwife with the study Project Director as a co-facilitator. At each of the visits participants will engage in self-assessments of weight and blood pressure, including learning to take their blood pressure with a digital cuff, calculating BMI, and plotting their weight gain on a graph), receive short individual clinical examinations from a midwife, and participate in group discussions about prenatal care, childbirth preparation, and their postpartum care. The session at 6-weeks postpartum will allow women to introduce their babies to the group and share childbirth stories.
  Arms: pregnant women receiving group prenatal care (GPNC)
Behavioral: Standard of Care — Standard of prenatal care
  Arms: pregnant women receiving standard of care (SOC)

SUMMARY:
To test the efficacy of a group prenatal care intervention to reduce the risk of obesity related health conditions during and after pregnancy in obese mothers and their infants.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility, acceptability, and preliminary efficacy of a group prenatal care (GPNC) intervention designed to reduce the risk for obesity related health conditions during and after pregnancy in overweight/obese mothers and their infants in American Samoa.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age. We will exclude younger pregnant women because adolescents may still be experiencing their own growth and development, which would be a source of confounding for our study outcomes.
* Self-reported Samoan ethnicity. Based on all four grandparents (of the participant) being reported as Samoa. Other ethnic groups make up approximately 2% of the American Samoan population but we are specifically interested in determining the efficacy of this intervention fro Samoan women, who have considerably poorer health outcomes in this setting.
* English speaking. The intervention will be delivered primarily in English, as is usual for standard prenatal care in this setting, with some Samoan language likely to be used in group discussions. Take home materials will be provided in both English and Samoan.
* Planning to reside in American Samoa for the duration of pregnancy and until at least 6 weeks postpartum. Some women travel from the neighboring country of Samoa (Independent/Western Samoa) to receive prenatal care at LBJTMC. These women will be excluded based on the need to receive all intervention sessions and a postpartum follow up.
* Singleton, viable pregnancy. A twin pregnancy reduced to singleton before 140 weeks by project gestational age is acceptable. An ultrasound must be conducted before randomization that shows a fetal heartbeat; there must be no evidence of more than one fetus on the most recent pre-randomization ultrasound. Including multiple pregnancies would confound study outcomes.
* Completed LBJTMC prenatal care enrollment visit. Participants must have enrolled in standard prenatal care and received a standard of care physical exam, ultrasound, confirmation of pregnancy dating, pregnancy history, and preliminary gestational diabetes screen to ensure that no pregnancy health-based exclusion criteria (see below) are met. Participants must obtain written documentation from their provider of this visit, and permission from them to participate in the GPNC study.
* Gestational age at randomization no earlier than 11 weeks 0 days and no later than 14 weeks 0 days based on an algorithm that compares the last menstrual period date and data from the enrollment ultrasound. This will ensure that each participant is exposed to the intervention for the same amount of time.
* Body mass index ≥ 26kg/m2 based on measured weight at enrollment and on measured height. The earliest weight measurement before randomization, measured specifically for the study will be used. A BMI cutpoint of 26 kg/m2 is used in line with the usual upward-adjusted criteria for overweight in populations of Polynesian descent.

Exclusion Criteria:

* Age less than 18 years because of the potential for growth during pregnancy and the need for participant informed consent.
* Diagnosis of diabetes prior to pregnancy or an HbA1C ≥ 6.5% or other glucose tolerance test result suggestive of pre-pregnancy diabetes. All potential participants will have HbA1C or an alternative test performed prior to randomization at their standard prenatal care enrollment visit.
* Gestational diabetes or preeclampsia in a previous pregnancy
* Known fetal anomaly/pregnancy health condition known to require specialist monitoring/treatment
* Planned termination of pregnancy
* Past history of anorexia or bulimia by medical history or patient report. Binge eating disorder (BED) is not an exclusion criterion.
* Current eating disorder diagnosed by a clinician
* Prior bariatric surgery
* Current use of one or more of the following medications:

  * Metformin
  * Systemic steroids
  * Antipsychotic agents (e.g. Abilify, Haldol, Risperdal, Seroquel, Zyprexa)
  * Anti-seizure medications or mood stabilizers that would be expected to have a significant impact on body weight (e.g Depakote, Lamictal, Lithium, Neurontin, Tegretol, Topamax, Keppra)
  * Medications for Attention Deficit Hyperactivity Disorder (ADHD) including amphetamines and methylphenidate
* Continued use of weight loss medication including Over The Counter (OTC) and dietary supplements for weight loss (e.g. Adipex, Suprenza, Tenuate, Xenical, Alli, conjugated linoleic acid, Hoodia, Green tea extract, Guar gum, Hydroxycut, Sensa, Corti-Slim, Chromium, Chitosan, Bitter Orange)
* Contraindications to aerobic exercise in pregnancy specified by the American College of Obstetrics and Gynocology (ACOG) committee Opinion #267, 2002 (re-affirmed 2009)
* Participation in another interventional study that influences weight control
* Participants unwillingness or inability to commit to a six-week postpartum follow up of herself or her child, including planning to move away
* Untreated medical or psychiatric condition (e.g. depression, bipolar disorder) that could impede study participation
* Hospitalization for hyperemesis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women of self-reported Samoan ethnicity.
Enrollment: 80 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
limiting weight gain | week 0
  initial weight measurement
limiting weight gain 0.5-0.7 lbs per week for overweight women | week 36 to week 40
  weight measurement
limiting weight gain 0.4-0.6 lbs per week for obese women | week 36 to week 40
  weight measurement
limiting weigh gain 0.4-0.6 lbs per week for obese women | 6 weeks postpartum
  weight measurement
limiting weigh gain 0.5-0.7 lbs per week for overweight women | 6 weeks postpartum
  weight measurement

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Hawley, PhD, Principal Investigator — Yale University